CLINICAL TRIAL: NCT05094531
Title: Implementation of a Post-traumatic Stress Disorder Primary Prevention Program Within the French Army
Brief Title: Implementation of a Post-traumatic Stress Disorder PREvention Program Within the French ARmy
Acronym: PREPAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Urgotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020PBMD03
Record Dates: First submitted 2021-04-26; First posted 2021-10-26 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Primary prevention programm; prevention; programm; Biopsychosocial; approach
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Masking Description: none since it is an open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants of this experimental group will have to attend the prevention program which is organised in eight 2-hour workshops, one every other week.
  Groups of 10-12 participants will be established prior to the first session of the program and will remain the same throughout the program.
  Interventions: Other: Primary prevention programm
- No-intervention group (No Intervention): Participants of the no-intervention group will not have to attend the prevention program.

INTERVENTIONS:
Other: Primary prevention programm — This programm aims to adress three dimensions : (i) biophysiology (flexibility of the autonomic nervous system), (ii) psychology (flexibility of coping strategies, sens of mission) and (iii) the social (stigmatization, seeking health care).
  Arms: Intervention group

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is a mental health condition that's triggered by a terrifying event perceived as a life threatening - either experiencing it or witnessing it. Lifetime prevalence of PTSD in the European population is between 0.7% and 1.9%. According to the "dose-response" model, the individuals most exposed to traumatic events (TEs) are those who are most at risk of developing this disorder. This is why it is not surprising to observe a higher prevalence of this disorder in the military population, ranging from 10% to 18% or even 45%, depending on the studies.

In the 1980s, the practice of evidence-based preventive medicine (EBM-Evidence Based Medicine) was developed. It involves the conscientious, explicit, judicious and reasonable use of modern, best evidence in making decisions about the care of individual patients. EBM integrates clinical experience and patient values with the best available research information. Health condition prevention includes several levels of action: primary, secondary or tertiary, depending on the timing of the intervention in the course of the disease.

The aim of this project is to explore the efficiency of primary prevention actions in strengthening the resilience capacities of at-risk professionals, such as the military, in order to prevent the development of PTSD and to improve it prognosis.

The objectives of this project are (i) to design a primary prevention program for PTSD specific to the military population studied and compatible with the operational constraints of field soldiers, (ii) then, to implement / validate it within the operational staff of the Mountain Infantry Brigade (MIB).

Our approach is based on an integrative reading of the processes in the risk of developing PTSD. This biopsychosocial approach targets both the factors specific to the individual (on the physiological and psychological level) and the contextual and social factors relating to his professional environment.

Three dimensions are addressed: (i) biophysiology (by integrating the study of key biomarkers of the neurobiological response to stress, and by strengthening the flexibility of the autonomic nervous system), (ii) psychology (by facilitating and measuring the development of the flexibility of coping strategies to cope with stress as well as by evaluating the moderating role of the sense mission in the development of PTSD) and (iii) the social (by facilitating community strategies aimed at reducing stigmatization and facilitating the use of care for professionals in difficulty in the institutional context).

ELIGIBILITY:
Inclusion Criteria:

* Social security affiliation
* Combat unit soldier with certificate of military efficiency
* With at least a 12-months employment contract within the MIB
* Able to attend all the workshops
* Not member of the Groupement Commando de Montagne

Exclusion Criteria:

* Participant of the PREPAR Phase 1
* Under chronic medication (daily treatment for at least a month)
* Unwilling to participate
* With a overseas deployment scheduled within the next 12 months
* Adult persons subject to a legal protection measure

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-05-29 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the prevention program in improving resilience at the end of the propgramm | After the completion of the programm, up to 50 weeks
  Composite primary endpoint. Significant improvement of resilience will be achieved if 2 or the following 3 criteria are meet:
  * 20% increase of the PANAS score (Positive And Negative Affect Schedule)
  * 20% score improvement of the SCS score (Self-Compassion Scale)
  * 5% score improvement of DRS-15 (Dispositional Resilience Scale)

SECONDARY OUTCOMES:
Follow-up evaluation of the resilience score | Two and six months after the completion of the prevention program
  Composite endpoint. Significant improvement of resilience will be achieved if 2 or the following 3 criteria are meet:
  * 20% increase of the PANAS score (Positive And Negative Affect Schedule)
  * 20% score improvement of the SCS score (Self-Compassion Scale)
  * 5% score improvement of DRS-15 (Dispositional Resilience Scale)

CONTACTS AND LOCATIONS:
Locations (1):
- 27 BIM, Varces-Allières-et-Risset, France

REFERENCES:
- [Derived] Le Barbenchon E, Trousselard M, Pellissier S, Moisseron-Baude M, Chachignon P, Bouny P, Toure Cuq E, Jacob S, Vigier C, Hidalgo M, Claverie D, Duffaud AM. Implementation of a Primary Prevention Program for Posttraumatic Stress Disorder in a Cohort of Professional Soldiers (PREPAR): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Jan 26;13:e47175. doi: 10.2196/47175. PMID 38277204